CLINICAL TRIAL: NCT00756457
Title: The Effect of Bracing and Strengthening Exercises on Posterior Tibial Tendon Dysfunction
Brief Title: Bracing and Strengthening for Posterior Tibial Tendon Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ithaca College (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R15AR054507 (NIH); R15AR054507 (NIH)
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Posterior Tibial Tendon Dysfunction
Keywords: PTTD; Tendinopathy; Tendon Injuries; Muscular Diseases; Foot Diseases
MeSH Terms: conditions — Posterior Tibial Tendon Dysfunction; Tendinopathy; Tendon Injuries; Muscular Diseases; Foot Diseases | interventions — Braces; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment Group (Active Comparator): Participants in Group A will undergo bracing and perform stretching exercises.
  Interventions: Device: Bracing; Other: Stretching exercises
- Passive Treatment Group (Experimental): Participants in Group B will undergo bracing and perform stretching and strengthening exercises.
  Interventions: Device: Bracing; Other: Strengthening exercises; Other: Stretching exercises

INTERVENTIONS:
Device: Bracing — Participants will wear a brace that includes ankle stirrup support and medial longitudinal arch support. The brace will be worn during weight-bearing tasks throughout the 12-week study.
  Other Names: Air Lift Brace
Other: Strengthening exercises — Participants performed strengthening exercises progressively longer each time for up to 3 sets of 30 repetitions twice daily by the third visit. Exercises included bilateral heel raises, foot adduction/rear foot inversion with thera-tubing, and unilateral heel raises. Participants increased resistance by using thera-bands with higher levels of resistance over the 12 week period. The amount of resistance was progressed according to patient tolerance at each visit. Strengthening exercises were preceded by the control stretching exercises which constituted a "warm up."
  Arms: Passive Treatment Group
Other: Stretching exercises — Subjects were provided with written descriptions and pictures demonstrating 2 range-of-motion exercises which included a wall calf stretch, and a supine ankle active range-of-motion exercise. Subjects were instructed to perform 3 sets of the stretching exercises, 2 times a day, similar to the intervention group. Each stretching exercise was performed twice and held for 30 seconds.

SUMMARY:
Posterior tibial tendon dysfunction (PTTD) is a problem with the tendon connecting one of the lower leg muscles to the foot bone. PTTD can cause pain, swelling, and a flattened foot and may require surgery if left untreated. Normal treatment for PTTD includes physical therapy exercise. In treating similar conditions in the lower leg, exercises that are active, like strengthening, seem to have better results than exercises that are passive, like stretching. This study will determine whether adding strengthening exercises to a normal PTTD treatment that includes wearing a brace and stretching is more beneficial than just wearing a brace and stretching.

DETAILED DESCRIPTION:
Posterior tibial tendon dysfunction (PTTD) involves inflammation, overstretching, or both of the posterial tibial tendon, which connects the tibialis posterior muscle to the bones in the foot. PTTD can cause pain in the inner ankle and development of a flat foot. Without treatment, correction of PTTD may require surgery. Standard interventions that may prevent the need for surgery include orthotic devices, bracing, and physical therapy, among other possibilities. Within physical therapy, foot exercises can be either active-as in the case of strengthening exercises-or passive-as in the case of stretching exercises. Evidence from clinical treatment of similar conditions suggests that active exercises are more effective than passive exercises in leading to recovery. This study will determine whether adding strengthening exercises to a normal intervention of bracing and stretching is more effective in improving a range of symptoms in stage II PTTD patients than using only bracing and stretching exercises.

Participants with Stage II PTTD will be recruited and placed in one of two groups for the duration of the 12-week study. The first group will undergo regular bracing and perform stretching exercises. The second group will undergo regular bracing and perform stretching and strengthening exercises. Braces, worn during weight-bearing tasks throughout the study, will include ankle stirrup support and medial longitudinal arch support. Strengthening exercises, which will be preceded by a warm-up of the posterior tibialis muscle, will include bilateral heel raises, foot adduction and rear foot inversion with thera-tubing, and unilateral heel raises. Frequency of exercise and number of repetitions will increase over the course of the study until participants are performing 3 sets of 30 repetitions 2 times per day. Assessments, which will occur at study entry, after 6 weeks, and after 12 weeks, will include foot range of motion, length of the posterior tibial muscle, and self-assessments of function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage II PTTD disorder
* Flexible flat foot deformity
* Palpable tenderness of posterior tibial tendon
* Swelling of the posterior tibial tendon sheath
* Pain during single limb heel rise
* Abnormal rear foot valgus
* Abnormal fore foot abduction as compared to contralateral side

Exclusion Criteria:

* Unable to walk for more than 15 meters
* Comorbidity within the foot
* Loss of protective sensation of the foot, as indicated by Semmes-Weinstein monofilament test of 5.07
* Inflammatory arthropathies
* Score greater than 23 on Mini Mental Status exam
* Arch index of less than 0.255
* Inability to assume a subtalar neutral posture
* PTTD in both feet

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff R. Houck, PhD, PT, Principal Investigator — Ithaca College - Rochester Center
Locations (1):
- Ithaca College - Rochester Center, Rochester, New York, United States

REFERENCES:
- [Derived] Houck J, Neville C, Tome J, Flemister A. Randomized Controlled Trial Comparing Orthosis Augmented by Either Stretching or Stretching and Strengthening for Stage II Tibialis Posterior Tendon Dysfunction. Foot Ankle Int. 2015 Sep;36(9):1006-16. doi: 10.1177/1071100715579906. Epub 2015 Apr 9. PMID 25857939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2007 - 2009 88 potential participants were screened from a university medical center.
Groups:
- Brace & Exercise: Participants in Group A will undergo bracing and perform stretching exercises.
- Brace: Participants in Group B will undergo bracing and perform stretching and strengthening exercises.
Period: Overall Study
Arm/Group | Brace & Exercise | Brace
Started | 20 | 19
Completed | 19 (One participant in the Active treatment group decided to have surgery after the 2 week follow-up.) | 17 (One participant moved overseas; the other participant resumed cancer treatment)
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brace & Exercise | Brace | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.9) | 58.1 (9.3) | 57.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Foot Function Index(FFI)
Description: The Foot Function Index (FFI) is a validated disease specific questionnaire that has been used to document outcomes in uncontrolled studies of PTTD. The domains of the 23 item FFI questionnaire include pain, disability, and activity limitations. The scale was originally validated in subjects with foot problems related to rheumatoid arthritis patients, and has subsequently been used to measure outcomes for a variety of foot and ankle problems including plantar fasciitis, diabetes, and PTTD. In clinical trials, the FFI has been used to detect change attributable to orthotics, plantar fasciitis, and brace use in PTTD. The three domains of the FFI include pain (FFI-Pain) range 0 to 90, disability (FFI-Disability) range 0- 90, and activity limitations (FFI-Activity Limitations) range 0 to 50. Each category asks patients to rate items relative to pain with higher scores indicating greater pain. The average of the three scales is the FFI-Total.
Time Frame: Measured at Weeks 1, 6, and 12
Population: A power analysis was performed based on previous a previous study. Only the participants that completed the study are included in the analysis. One participant opted to have surgery at 2 weeks from the Brace & Exercise group. One participant moved overseas and the other resumed cancer treatments bringing the total to 17.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Brace & Exercise (Baseline); Brace & Exercise (6 Weeks); Brace & Exercise (12 Weeks): This group based on the inclusion exclusion criteria were classified as stage II PTTD.
- Brace (Baseline); Brace (6 Weeks); Brace (12 Weeks): This group based on the inclusion and exclusion criteria was classified as having stage II PTTD.
Arm/Group | Brace & Exercise (Baseline) | Brace (Baseline) | Brace & Exercise (6 Weeks) | Brace (6 Weeks) | Brace & Exercise (12 Weeks) | Brace (12 Weeks)
Number analyzed (Participants) | 19 | 17 | 19 | 17 | 19 | 17
units on a scale
  FFI - Activity Limitation (range 0 - 30) | 16.0 (11.2) | 12.7 (12.0) | 8.1 (8.6) | 8.3 (8.9) | 9.8 (12.6) | 6.7 (7.3)
  FFI - Disability (range 0 - 90) | 40.0 (20.4) | 30.6 (15.4) | 21.3 (14.6) | 20.8 (13.1) | 24.4 (21.6) | 17.8 (13.5)
  FFI- Pain (range 0 - 50) | 37.5 (18.4) | 34.6 (11.6) | 20.6 (14.5) | 21.2 (14.0) | 19.1 (17.4) | 18.4 (13.8)
  FFI - Total | 31.2 (13.2) | 26.0 (10.6) | 16.7 (11.5) | 16.8 (10.1) | 17.8 (15.9) | 14.3 (10.1)

2. Secondary Outcome: Foot Kinematics and Posterior Tibial Muscle Length (Estimated From Foot Kinematics)
Description: A 3 dimensional foot kinematic model including the tibia, calcaneus (hindfoot), 1st metatarsal, 2-4th metatarsals and hallux was used to measure foot movement. Six infrared cameras (Optotrak Motion Analysis System, Northern Digital Inc, CAN), synchronized with force plate data (Model 9286, Kistler, Switzerland), were used to collect kinematics (60 Hz) and force (1000 Hz) data with the Motion Monitor software Version 7.24 (Motion Monitor, Innsport Training Inc, USA). Anatomically based coordinate systems were established for each segment using digitized boney landmarks consistent with a previous study. Kinematic data were smoothed using a 4th order, zero phase lag, Butterworth filter with a cut off frequency of 6 Hz. To calculate relative joint angles a Cardan angle Z-X-Y sequence of rotations was used as suggested by Cole et al. The range of possible values varies for each individual and each joint.
Time Frame: Measured at Weeks 1,6 and 12
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Brace & Exercise (Baseline); Brace & Exercise (6 Weeks); Brace & Exercise (12 Weeks): This group based on the inclusion and exclusion criteria was classified as having stage II PTTD. Only the participants that completed the study are included here. One participant opted to have surgery after 2 weeks of treatment.
- Brace (Baseline); Brace (6 Weeks); Brace (12 Weeks): This group based on the inclusion and exclusion criteria was classified as having stage II PTTD. Only the participants that completed the study are included here. One participant moved overseas and another resumed cancer treatments bringing the total to 17.
Arm/Group | Brace & Exercise (Baseline) | Brace (Baseline) | Brace & Exercise (6 Weeks) | Brace (6 Weeks) | Brace & Exercise (12 Weeks) | Brace (12 Weeks)
Number analyzed (Participants) | 19 | 17 | 19 | 17 | 19 | 17
Degrees
  Hindfoot In(+)/Ev(-) (5% Stance) | -8.6 (3.2) | -8.8 (3.8) | -8.4 (3.1) | -8.2 (3.7) | -8.7 (2.8) | -8.8 (4.0)
  Hindfoot In(+)/Ev(-) (39% Stance) | -10.8 (2.4) | -10.6 (3.0) | -11.2 (2.9) | -10.2 (3.6) | -10.5 (3.1) | -10.6 (3.4)
  Hindfoot In(+)/Ev(-) (84% Stance) | -4.9 (3.7) | -4.2 (3.5) | -5.5 (3.1) | -4.6 (3.6) | -4.5 (4.4) | -4.5 (3.9)
  Hindfoot Df(+)/Pf(-) (5% Stance) | -8.8 (3.6) | -7.5 (3.3) | -3.4 (4.6) | -0.4 (5.6) | -4.0 (4.8) | -1.0 (6.3)
  Hindfoot Df(+)/Pf(-) (39% Stance) | 0.2 (2.9) | 2.4 (3.8) | 6.2 (3.7) | 9.7 (4.8) | 6.3 (4.3) | 9.1 (6.4)
  Hindfoot Df(+)/Pf(-) (84% Stance) | 5.7 (4.3) | 6.8 (4.6) | 11.9 (5.4) | 14.0 (7.3) | 11.8 (4.6) | 13.6 (7.7)
  1st Met Ad(+)/Ab(-) (5% Stance) | -6.5 (3.2) | -7.2 (3.2) | -6.3 (3.2) | -7.4 (2.6) | -6.4 (2.9) | -6.7 (3.2)
  1st Met Ad(+)/Ab(-) (39% Stance) | -5.2 (3.3) | -6.9 (2.5) | -5.1 (3.0) | -6.9 (2.3) | -5.2 (2.6) | -6.4 (2.9)
  1st Met Ad(+)/Ab(-) (84% Stance) | -6.7 (4.9) | -7.4 (4.2) | -6.6 (5.0) | -7.5 (4.0) | -7.5 (4.5) | -7.4 (4.3)
  1st Met Df(+)/Pf(-) (5% Stance) | 11.2 (6.5) | 8.2 (6.1) | 11.4 (6.5) | 8.5 (7.0) | 12.6 (7.1) | 9.1 (6.4)
  1st Met Df(+)/Pf(-) (39% Stance) | 14.8 (6.1) | 11.7 (5.7) | 14.3 (5.9) | 11.9 (6.3) | 15.6 (6.3) | 12.6 (5.5)
  1st Met Df(+)/Pf(-) (84% Stance) | 14.2 (8.6) | 12.6 (6.9) | 14.2 (7.7) | 12.4 (8.3) | 14.8 (8.3) | 13.3 (7.3)

3. Primary Outcome: Short Musculoskeletal Functional Assessment
Description: The Short Musculoskeletal Function Assessment Questionnaire (SMFA) is a 46 item self-report questionnaire consisting of the Dysfunction Index, which has thirty-four items, and the Bother index which has 12 items. The Dysfunction index is used for assessment of patient perceptions of functional performance while the Bother index is used to assess patients' perceptions of the degree patients are bothered in broad areas such as recreation and leisure. The responsiveness to change of the SMFA is 10 points out a range of 100 for each scale (Dysfunction, Mobility, and Bother indexes). The SMFA is also particularly suitable for the current investigation due to the presence of a sub-category of questions from the Dysfunction Index that pertains specifically to mobility (i.e. Mobility Index). Lower scores (lowest = 0) indicate better function, mobility, and that patients are less bothered while higher scores (highest = 100) indicate worse function, mobility and that patients are bothered.
Time Frame: Measured at Weeks 1, 6, and 12
Measure: Mean (Standard Deviation); unit: score
Groups:
- Brace (Baseline); Brace (6 Weeks); Brace (12 Weeks): This group based on the inclusion and exclusion criteria was classified as having stage II PTTD. Only the participants that completed the study are included here. One participant moved overseas and the other resumed cancer treatments bringing the total to 17.
Arm/Group | Brace & Exercise (Baseline) | Brace (Baseline) | Brace & Exercise (6 Weeks) | Brace (6 Weeks) | Brace & Exercise (12 Weeks) | Brace (12 Weeks)
Number analyzed (Participants) | 19 | 17 | 19 | 17 | 19 | 17
score
  Dysfunction (Range 0- 100) | 22.2 (12.3) | 16.6 (9.0) | 13.0 (9.1) | 12.9 (7.2) | 14.5 (9.1) | 11.7 (6.3)
  Mobility (Range 0 - 100) | 26.6 (14.2) | 22.1 (11.6) | 15.2 (10.6) | 18.4 (10.6) | 17.0 (10.7) | 15.5 (8.2)
  Bother (Range 0 - 100) | 25.8 (20.1) | 22.8 (16.4) | 15.1 (13.9) | 13.7 (9.2) | 16.4 (18.9) | 11.8 (6.4)

4. Secondary Outcome: Foot Strength
Description: A force transducer (Model SML-200, Interface, Scottsdale, AZ) was connected in series with a resistance plate and oscilloscope (TDS 410A, Tektronix, Beaverton, OR) to display force readings. Participants were seated with their leg in an an air stirrup brace (Aircast, Inc.) mounted on uprights. The air stirrup brace was adjusted so the heel was approximately 10 cm above the resistance plate, resulting in 30 to 45 degrees of ankle plantar flexion depending on foot length. The resistance plate was mounted on ball bearing tracks in the medial/lateral direction and moleskin was used to fit to the general shape of the medial forefoot. The result was that participants could exert maximum effort against the resistance plate (medial direction) with little discomfort. This testing position essentially replicates the manual muscle test position for the posterior tibialis muscle. Force in Newtons was then divided by body mass in kilograms to calculate normalized strength (N/Kg).
Time Frame: Measured at Weeks 1, 6, and 12
Measure: Mean (Standard Deviation); unit: N/kg
Groups:
- Brace & Exercise (Baseline); Brace & Exercise (6 Weeks); Brace & Exercise (12 Weeks): This group based on the inclusion and exclusion criteria was classified as having stage II PTTD. Only the participants that completed the study are included here. One participant opted to have surgery after 2 weeks of treatment bringing the total to 19.
Arm/Group | Brace & Exercise (Baseline) | Brace (Baseline) | Brace & Exercise (6 Weeks) | Brace (6 Weeks) | Brace & Exercise (12 Weeks) | Brace (12 Weeks)
Number analyzed (Participants) | 19 | 17 | 19 | 17 | 19 | 17
N/kg
  Involved Subtalar Inversion Strength | 0.70 (0.20) | 0.79 (0.25) | 0.77 (0.21) | 0.86 (0.29) | 0.78 (0.21) | 0.82 (0.25)
  Uninvolved Subtalar Inversion Strength | 0.81 (0.16) | 0.94 (0.25) | 0.84 (0.18) | 0.99 (0.22) | 0.85 (0.13) | 0.99 (0.23)

ADVERSE EVENTS:
Time Frame: The study period monitored participants for12 weeks. Adverse events were recorded at 1, 6 and 12 weeks.
Arm/Group | Brace & Exercise | Brace
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No